CLINICAL TRIAL: NCT01436240
Title: Linguistic Validation of the Spanish Translation of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Brief Title: Spanish Translation of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ralph Lauren Center for Cancer Care and Prevention (Other); M.D. Anderson Cancer Center (Other); St. Joseph's Hospital, Los Angeles (Unknown); Hektoen Stroger Hospital (Unknown); University of Miami (Other); National Cancer Institute (NCI) (NIH); FACITtrans, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 11-133
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: Patient-Reported Outcomes; Common Terminology Criteria for Adverse Events; PRO-CTCAE; Native Spanish Speaking; Spanish Translation; Cognitive Interview; Questionnaire; 11-133; Adverse Events; chemotherapy; radiation therapy; treatment in previous 6 months
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Spanish-speaking Latino participants: The investigators will conduct up to two rounds of PRO-CTCAE (patient-reported outcome- Common Terminology Criteria for Adverse Events) version questionnaire administration followed by cognitive interviews in Spanish-speaking Latino patients who are receiving cancer treatment or who have completed treatment for cancer within the past six months at one of the participating sites.
  Interventions: Behavioral: questionnaire administration followed by cognitive interviews

INTERVENTIONS:
Behavioral: questionnaire administration followed by cognitive interviews — Each cognitive interviewing procedure will include two parts. Participants will first be asked to independently complete a series of PRO-CTCAE symptom items in a Patient Questionnaire. Following completion by the participant of the Patient Questionnaire containing PRO-CTCAE items, the bilingual interviewer will query participants regarding item comprehension, relevance, inclusiveness, cultural appropriateness, and cognitive processes used to generate responses, via a semi-scripted cognitive debriefing interview developed to assure consistency across interviews.

SUMMARY:
The purpose of this study is to see if questions in English about symptoms that patients may have during cancer treatment are understandable when translated into Spanish. These questions will later be used in future studies to give a better understanding of patient symptoms".

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older and be able to provide informed consent.
* Participants must be patients being followed for clinical care at one of the collaborating sites, and must be either currently undergoing or having completed treatment (chemotherapy or radiation therapy) for cancer in the previous 6 months.
* Participants must be native Spanish-speakers.
* Participants must be able either to read and understand the items in Spanish or to hear and understand and respond to the items when read to them verbatim in Spanish.

Exclusion Criteria:

* Cognitive impairment as determined by the patient's Physician or Nurse which or study coordinators renders them unable to understand the items or report on his/her symptoms from the last 7 days.
* Participants who have only received surgery are not eligible
* If participants request to have the consent form in English, they will not be eligible for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited from five different collaborating sites: MSKCC/Ralph Lauren Center for Cancer Care and Prevention, MD Anderson, University of Miami, Stroger Hospital, and St. Joseph's Hospital. Approximately 40 participants will be enrolled at MSKCC; 120 participants will be enrolled in total.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
the ability for the PRO-CTCAE system to be used in Spanish-speaking populations in the U.S. | 2 years
  Patient Questionnaire (either via paper or read to them verbatim), and undergo a subsequent cognitive interview, as described in this protocol. Interviews will be conducted either by bilingual site staff who have been trained to conduct these interviews, or by trained bilingual interviewers from FACITtrans

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Basch, MD, MSc, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - St Joseph'S Hospital, Los Angeles, California
  - University of Miami, Miami, Florida
  - Hektoen /Stroger Hospital, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Arnold B, Mitchell SA, Lent L, Mendoza TR, Rogak LJ, Barragan NM, Willis G, Medina M, Lechner S, Penedo FJ, Harness JK, Basch EM; PRO-CTCAE Spanish Translation and Linguistic Validation Study Group. Linguistic validation of the Spanish version of the National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Support Care Cancer. 2016 Jul;24(7):2843-51. doi: 10.1007/s00520-015-3062-5. Epub 2016 Feb 2. PMID 26838022
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm